CLINICAL TRIAL: NCT00120900
Title: A Phase III, 12-week, Multicentre, Double-Blind, Double-Dummy, Randomised, Placebo - and Active Comparator - Contolled, Parallel Group Study to Investigate the Efficacy and Safety of GW406381 XXmg and YYmg Administered Orally Once Daily, in Adults With Osteoarthritis of the Knee
Brief Title: Evaluation of GW406381 in Treating Adults With Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXA30007
Record Dates: First submitted 2005-06-30; First posted 2005-07-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis, Knee
Keywords: COX-2 inhibitor; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — GW406381X

INTERVENTIONS:
Drug: GW406381

SUMMARY:
This study was designed to evaluate the effectiveness of GW406381 (a COX-2 inhibitor) in treating the signs and symptoms of osteoarthritis of the knee.

DETAILED DESCRIPTION:
A Phase III, 12-week, Multicentre, Double-blind, Double-dummy, Randomised, Placebo- and Active Comparator-Controlled, Parallel Group study to investigate the Efficacy and Safety of GW406381 1mg, 5mg, 10mg, 25mg and 50mg administered orally once daily, in adults with Osteoarthritis of the knee (CXA30007).

ELIGIBILITY:
Inclusion criteria:

* Subjects have a primary diagnosis of osteoarthritis of the knee with symptom duration of at least 3 months.
* Use pain medication, such as a COX-2 inhibitor or NSAID (non-steroidal anti-inflammatory drug) at least 5 days per week.

Exclusion criteria:

* History of hypersensitivity or intolerance to pain medications.
* History of gastroduodenal perforations and/or obstructions.
* History of upper GI (gastrointestinal) ulceration within the previous 6 months.
* History of upper or lower GI bleeding within the previous year.
* History of inflammatory bowel disease.
* Currently take sucralfate or misoprostol.
* Currently taking aspirin daily for the heart.
* Other restrictions around the use medications apply and would need to be discussed.
* History of coronary artery disease, (angina, MI) or surgery.
* History of congestive heart failure or renal artery stenosis.
* History of stroke or transient ischemic attack.
* History of uncontrolled hypertension.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1340 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in OA symptoms at week 12 as measured by scores on subject-completed questionnaires on pain, daily activities and global assessment

SECONDARY OUTCOMES:
Change in OA symptoms as measured by subject and physician-completed questionnaires at each scheduled visit. Percentage of responders, subjects discontinuing due to lack of efficacy, use of rescue medication and health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- GSK Investigational Site, Ishøj, Denmark
- Netherlands (3):
  - GSK Investigational Site, De Bilt
  - GSK Investigational Site, Ewijk
  - GSK Investigational Site, Heerlen
- Norway (5):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Hønefoss
  - GSK Investigational Site, Lier
  - GSK Investigational Site, Oslo
- South Korea (3):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
- GSK Investigational Site, San Juan, Spain
- GSK Investigational Site, Helsingborg, Sweden